CLINICAL TRIAL: NCT03138317
Title: Evaluation of Platelet Rich Plasma (PRP) for Knee Osteoarthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: RDO Laboratory (Unknown)
Responsible Party: Principal Investigator, Ricardo Fuller, Assistant of Osteoarthritis ambulatory; PhD researcher., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2017-04-16; First posted 2017-05-03 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP (Experimental): Goup 1: knee injection of Platelet Rich Plasma (PRP)
  Interventions: Biological: PRP
- Plasma (Experimental): Group 2: knee injection of Plasma
  Interventions: Biological: Plasma
- Placebo (Placebo Comparator): Group 3: knee injection of placebo (saline solution)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PRP — This group will receive a knee injection with 6 ml of platelet rich plasma (PRP)
  Arms: PRP
Biological: Plasma — This group will receive a knee injection with 6 ml of plasma.
  Arms: Plasma
Biological: Placebo — This group will receive a knee injection with 6 ml saline solution.
  Arms: Placebo

SUMMARY:
Study was designed to evaluate efficacy of autologous platelet rich plasma (PRP) injections guided by ultrasound for treatment of knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most prevalent rheumatic disease in the world and its treatment is still relatively limited. The efficacy of platelet rich plasma (PRP) for treatment of osteoarthritis of knees has been demonstrated both in vitro and in vivo. Numerous studies published in literature show a good potential of PRP in treatment of osteoarthritis. However, results are not yet consistent due to methodological gaps such as lack of control, inadequate controls, inadequate assessment tools, inadequate matching for interventions, insufficient description of design and way of obtaining PRP.

The aim of the study is to evaluate efficacy of autologous PRP injections guided by ultrasound for treatment of knee osteoarthritis.

Patients will be randomized into three groups for ultrasound guided knee infiltrations: the first group will receive PRP, the second group will receive plasma and the third group will receive a placebo of physiological solution. All patients will be assessed using Visual Analog Pain Scale, WOMAC (Western Ontario McMasters University Osteoarthritis Index), Knee Injury and Osteoarthritis Outcome Score, conventional radiography, ultrasonography, and follow the standardization of results for clinical trials in Osteoarthritis (OMERACT-OARSI). Patients will be evaluated during clinical follow-up after 1, 4, 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged from 45 to 80 years
2. Fulfill criteria for knee osteoarthritis of the ACR - American College of Rheumatology (Altman et al., 1986)
3. Radiographic classification 2 or 3 by Kellgren and Lawrence score
4. Relate pain in the last week of 3 to 8 points on the Visual Analogue Scale - EVA (Bellamy et al., 1988)

Exclusion Criteria:

1. Use of analgesics, NSAIDs and myorelaxants less than a week before the start of the study.
2. Use of slow-acting drugs in osteoarthritis started less than 8 weeks before the start of the study. For cases that they have been in use for more than 8 weeks, they should be maintained until the end of the week.
3. Infiltration of corticosteroid or infiltration with hyaluronic acid in the six months prior to the start of the study.
4. Intra-articular infiltration with any medication in any other joint less than 1 month after inclusion;
5. Introduction of any medical or physiotherapeutic intervention in the last 3 months (rehabilitation, acupuncture, cane, orthotics, etc.) for locomotor system;
6. Body Mass Index (BMI) greater than 35.
7. Presence of other types of arthropathies such as rheumatoid arthritis, diffuse connective tissue diseases, microcrystalline arthropathies, spondyloarthropathies and infectious arthropathies.
8. Symptomatic osteoarthritis of hip and feet
9. Presence of known meniscal or symptomatic ligament damage in the studied knee;
10. Previous surgery in the studied knee.
11. Difference in length in lower limbs greater than 1 cm.
12. Presence of cutaneous lesion on the surface of the joint studied;
13. Important scoliosis.
14. Blood dyscrasia or use of anticoagulant;
15. Presence of other diseases: severe depression, diabetes, coagulopathies, decompensated cardiovascular disease, infection, immunosuppression (allowed MTX up to 10 mg), systemic infectious disease, symptomatic lower limb vascular disease, neurological diseases, neoplasia or any other conditions that may compromise the procedure in doctor evaluation;
16. To be receiving pension benefit due to osteoarthritis of the knees.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Knee pain score measured by Visual Analogue Scale (VAS) | 24 weeks
  Knee pain score measured by Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Dorio M, Pereira RMR, Luz AGB, Deveza LA, de Oliveira RM, Fuller R. Efficacy of platelet-rich plasma and plasma for symptomatic treatment of knee osteoarthritis: a double-blinded placebo-controlled randomized clinical trial. BMC Musculoskelet Disord. 2021 Sep 24;22(1):822. doi: 10.1186/s12891-021-04706-7. PMID 34560869